CLINICAL TRIAL: NCT06227689
Title: Evaluation of Vaccine Chatbot on HPV Vaccine Awareness and Vaccination for Middle School Girls in China: a Randomized Controlled Trial and Implementation Science Study
Brief Title: Effectiveness of Vaccine Chatbot on HPV Vaccine Awareness and Vaccination in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhiyuan Hou, Associate Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FudanU-HPV Chatbot
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: HPV Vaccine
Keywords: HPV vaccine; awareness; knowledge; vaccination; vaccine confidence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Chatbot Intervention group (Experimental): In this arm, participants will receive a vaccine chatbot intervention. They will be invited to use the HPV vaccine chatbot online through WeChat or any web browsers, where they can ask any questions related to the HPV vaccine and get immediate answers from the chatbot. The intervention lasts two weeks, with invitations sent every four days to reinforce the intervention.
  Interventions: Other: Vaccine chatbot that offering HPV vaccine-related information
- Control group (No Intervention): The control group will not use the chatbot during the intervention duration.

INTERVENTIONS:
Other: Vaccine chatbot that offering HPV vaccine-related information — The intervention group will be invited to use the HPV vaccine chatbot online through WeChat or any web browsers, where they can ask any questions related to the HPV vaccine and get previously validated answers from the chatbot immediately. All the answers will be drawn from a database, whose content were obtained from official websites of Chinese government, HPV vaccine enterprises, and International organizations like WHO, and had been validated by experts. The intervention lasts two weeks, with invitations sent every four days to reinforce the intervention.
  Arms: HPV Chatbot Intervention group

SUMMARY:
This interventional study targets female students in junior middle school. It goal is to evaluate the effectiveness of a vaccine chatbot on HPV vaccine awareness and vaccination. The main questions it aims to answer are:

1. How will the novel digital tool, a vaccine chatbot, impact eligible parents' awareness and knowledge of HPV vaccines, their willingness to vaccinate their daughters, and vaccination status of female students.
2. How is the vaccine chatbots accepted by all stakeholders, and what are the facilitators of and barriers to implementing vaccine chatbot promotion campaign.

The intervention group will go through the intervention measure while the control group will not:

1. The intervention group will be invited to use the HPV vaccine chatbot online through WeChat , the mostly widely used social media platform in mainland China, or any web browsers. They can ask any questions related to the HPV vaccine and get validated answers from the chatbot immediately. The intervention lasts two weeks, with invitations sent every four days to reinforce the intervention.
2. The control group will not use the chatbot during the intervention duration.

Researchers will compare participants' HPV vaccine awareness, and vaccination intention and status after intervention between intervention group and control group to evaluate if the vaccine chatbot improves HPV vaccine awareness and vaccination.

DETAILED DESCRIPTION:
This is a cluster randomized trial consisted of 2 arms to evaluate the effectiveness of a vaccine chatbot on parents' HPV vaccine awareness, knowledge, and vaccination intention and status regarding their daughters in junior middle school.

The sample size was calculated based on the primary outcome, which is the HPV vaccination rate among middle school girls, and the main analysis method, which involves comparing differences in rates or means before and after the intervention. According to a literature review, the current HPV vaccination rate among female students is around 5%. The investigators assumed that the vaccination rate could increase to between 10% and 12% following the intervention. The minimum sample size was calculated to be between 369 and 648 participants in each group, with a significance level (α) of 0.05, a test power (1-β) of 0.8, and a cluster design effect (D) of 1.5.

Multi-stage sampling will be employed. Firstly, three representative cities will be selected to represent the megacity, general urban city, and rural counties in China, respectively. Then, within each city, three or four middle schools will be selected based on economic development, school size, geographical location. Next, around six classes will be randomly selected for each of the three grades in each middle school. For all the female students who have not be vaccinated against HPV in selected classes, one of their parents will be included in the study. A total of around 162 classes are expected to be included, with around 54 classes in each city.

Stratified cluster randomized grouping will be employed. All classes will be grouped into intervention group or control group by class at a 1:1 ratio, stratified by city, school, and grades, resulting with around 81 classes into the intervention group and 81 in control group. Approximately 600 parents (300 in intervention group; 300 in control group) are expected to participate in the study in each city, with a total sample size of 1,800 parents, meeting the sample size requirement.

Baseline survey will be conducted before the intervention. Then, the intervention group will be invited to use the HPV vaccine chatbot online through WeChat or any web browsers, where they can ask any questions related to the HPV vaccine and get validated answers from the chatbot immediately. The intervention lasts two weeks, with invitations sent every four days to reinforce the intervention. The control group will not use the chatbot during the intervention duration. After 2 weeks, follow-up survey will then be conducted. HPV vaccination status of female students will be collected after 4 months.

The Generalized Estimating Equations (GEE) and mixed-effects analysis methods were employed to control for the effects of covariates and evaluate the intervention effect of the chatbot.

Besides impact evaluation, this study will also conduct an implementation science study, using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) framework to comprehensively assess the cost-effectiveness, applicability, and scalability of the HPV vaccine chatbot intervention in real-world. Both quantitative and qualitative methods will be used to evaluate its implementation across the above-mentioned five dimensions: reach, effectiveness, adoption, implementation, and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Parents of female students in middle school;
* The students not vaccinated or appointed for HPV vaccination and without contraindications to HPV vaccines;
* Without mental disorders or visual/reading impairments, and able to cooperate with and undergo the intervention activities;
* Obtained informed consent and willing to participate in the study.

Exclusion Criteria:

* Students vaccinated or appointed for HPV vaccination or with any contraindication to HPV vaccines;
* With mental disorders or visual/reading impairments, and unable to cooperate with and undergo the intervention activities;
* Unwilling to participate.

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccination status and appointment | Two weeks and four months after the baseline
  whether participants' daughters get vaccinated against HPV or have an appointment for vaccination, measured by self-report and validated by vaccination information system

SECONDARY OUTCOMES:
Willingness to vaccinate | Two weeks between baseline and follow-up surveys
  Parents' willingness to vaccinate their daughters against HPV, measured using a five-point Likert scale from "very unwilling" to "very willing"
HPV vaccine awareness and knowledge | Two weeks between baseline and follow-up surveys
  10 questions about HPV vaccine knowledge and misinformation. Total knowledge score is calculated based on the number of questions answered correctly by the participants.
HPV vaccine confidence | Two weeks between baseline and follow-up surveys
  Vaccine Confidence Index (VCI), including confidence on vaccine importance, effectiveness and safety
Healthcare consultation | Two weeks after the baseline
  Assessment of parental engagement in seeking medical advice about vaccinating their daughter with the HPV vaccine during the two weeks leading up to the follow-up survey.
Chatbot Usability | Two weeks after the baseline
  17 questions assessing usability and feasibility, fairness and safety, user experience, and overall assessment of the chatbot.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Hou, PhD, Principal Investigator — School of Public Health，Fudan University; Leesa Lin, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (2):
- China (2):
  - Chizhou Health Center for Disease Control and Prevention, Chizhou, Anhui
  - Jiading District Center for Disease Control and Prevention, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared upon reasonable requests. A written data-sharing request for meta-analysis should be submitted by email with a methodologically sound proposal. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta-analysis. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Hu S, Xu X, Zhang Y, Liu Y, Yang C, Wang Y, Wang Y, Yu Y, Hong Y, Zhang X, Bian R, Cao X, Xu L, Zhao F. A nationwide post-marketing survey of knowledge, attitude and practice toward human papillomavirus vaccine in general population: Implications for vaccine roll-out in mainland China. Vaccine. 2021 Jan 3;39(1):35-44. doi: 10.1016/j.vaccine.2020.11.029. Epub 2020 Nov 23. PMID 33243631
- [Result] Falcaro M, Castanon A, Ndlela B, Checchi M, Soldan K, Lopez-Bernal J, Elliss-Brookes L, Sasieni P. The effects of the national HPV vaccination programme in England, UK, on cervical cancer and grade 3 cervical intraepithelial neoplasia incidence: a register-based observational study. Lancet. 2021 Dec 4;398(10316):2084-2092. doi: 10.1016/S0140-6736(21)02178-4. Epub 2021 Nov 3. PMID 34741816
- [Result] Drolet M, Benard E, Perez N, Brisson M; HPV Vaccination Impact Study Group. Population-level impact and herd effects following the introduction of human papillomavirus vaccination programmes: updated systematic review and meta-analysis. Lancet. 2019 Aug 10;394(10197):497-509. doi: 10.1016/S0140-6736(19)30298-3. Epub 2019 Jun 26. PMID 31255301
- [Result] Sonawane K, Zhu Y, Montealegre JR, Lairson DR, Bauer C, McGee LU, Giuliano AR, Deshmukh AA. Parental intent to initiate and complete the human papillomavirus vaccine series in the USA: a nationwide, cross-sectional survey. Lancet Public Health. 2020 Sep;5(9):e484-e492. doi: 10.1016/S2468-2667(20)30139-0. Epub 2020 Jul 21. PMID 32707126
- [Result] Zang S, Zhang X, Qu Z, Chen X, Hou Z. Promote COVID-19 Vaccination for Older Adults in China. China CDC Wkly. 2022 Sep 16;4(37):832-834. doi: 10.46234/ccdcw2022.173. No abstract available. PMID 36284538
- [Result] Zhang Y, Wang Y, Liu L, Fan Y, Liu Z, Wang Y, Nie S. Awareness and knowledge about human papillomavirus vaccination and its acceptance in China: a meta-analysis of 58 observational studies. BMC Public Health. 2016 Mar 3;16:216. doi: 10.1186/s12889-016-2873-8. PMID 26936076
- [Result] Xie Y, Su LY, Wang F, Tang HY, Yang QG, Liu YJ. Awareness regarding and vaccines acceptability of human papillomavirus among parents of middle school students in Zunyi, Southwest China. Hum Vaccin Immunother. 2021 Nov 2;17(11):4406-4411. doi: 10.1080/21645515.2021.1951931. Epub 2021 Jul 29. PMID 34324411
- [Result] Wei Z, Liu Y, Zhang L, Sun X, Jiang Q, Li Z, Wu Y, Fu C. Stages of HPV Vaccine Hesitancy Among Guardians of Female Secondary School Students in China. J Adolesc Health. 2023 Jan;72(1):73-79. doi: 10.1016/j.jadohealth.2022.08.027. Epub 2022 Oct 11. PMID 36229401
- [Result] Zhang X, Wang Z, Ren Z, Li Z, Ma W, Gao X, Zhang R, Qiao Y, Li J. HPV vaccine acceptability and willingness-related factors among Chinese adolescents: a nation-wide study. Hum Vaccin Immunother. 2021 Apr 3;17(4):1025-1032. doi: 10.1080/21645515.2020.1812314. Epub 2020 Oct 29. PMID 33121330
- [Result] Zhang X, Liu CR, Wang ZZ, Ren ZF, Feng XX, Ma W, Gao XH, Zhang R, Brown MD, Qiao YL, Geng Q, Li J. Effect of a school-based educational intervention on HPV and HPV vaccine knowledge and willingness to be vaccinated among Chinese adolescents : a multi-center intervention follow-up study. Vaccine. 2020 Apr 29;38(20):3665-3670. doi: 10.1016/j.vaccine.2020.03.032. Epub 2020 Mar 31. PMID 32245644
- [Result] Wang D, Wu J, Du J, Ong H, Tang B, Dozier M, Weller D, Campbell C. Acceptability of and barriers to human papillomavirus vaccination in China: A systematic review of the Chinese and English scientific literature. Eur J Cancer Care (Engl). 2022 May;31(3):e13566. doi: 10.1111/ecc.13566. Epub 2022 Mar 1. PMID 35229931
- [Result] Si M, Su X, Jiang Y, Wang W, Zhang X, Gu X, Ma L, Li J, Zhang S, Ren Z, Liu Y, Qiao Y. Effect of an IMB Model-Based Education on the Acceptability of HPV Vaccination Among College Girls in Mainland China: A Cluster RCT. Cancer Control. 2022 Jan-Dec;29:10732748211070719. doi: 10.1177/10732748211070719. PMID 35088609
- [Result] Si M, Su X, Jiang Y, Wang W, Zhang X, Gu X, Ma L, Li J, Zhang S, Ren Z, Liu Y, Qiao Y. An Internet-Based Education Program for Human Papillomavirus Vaccination Among Female College Students in Mainland China: Application of the Information-Motivation-Behavioral Skills Model in a Cluster Randomized Trial. J Med Internet Res. 2022 Sep 30;24(9):e37848. doi: 10.2196/37848. PMID 36178723
- [Result] Luk TT, Lui JHT, Wang MP. Efficacy, Usability, and Acceptability of a Chatbot for Promoting COVID-19 Vaccination in Unvaccinated or Booster-Hesitant Young Adults: Pre-Post Pilot Study. J Med Internet Res. 2022 Oct 4;24(10):e39063. doi: 10.2196/39063. PMID 36179132
- [Result] Lee KY, Dabak SV, Kong VH, Park M, Kwok SLL, Silzle M, Rachatan C, Cook A, Passanante A, Pertwee E, Wu Z, Elkin JA, Larson HJ, Lau EHY, Leung K, Wu JT, Lin L. Effectiveness of chatbots on COVID vaccine confidence and acceptance in Thailand, Hong Kong, and Singapore. NPJ Digit Med. 2023 May 25;6(1):96. doi: 10.1038/s41746-023-00843-6. PMID 37231110
- [Result] Wilson L, Marasoiu M. The Development and Use of Chatbots in Public Health: Scoping Review. JMIR Hum Factors. 2022 Oct 5;9(4):e35882. doi: 10.2196/35882. PMID 36197708
- [Result] Almalki M, Azeez F. Health Chatbots for Fighting COVID-19: a Scoping Review. Acta Inform Med. 2020 Dec;28(4):241-247. doi: 10.5455/aim.2020.28.241-247. PMID 33627924
- [Result] Kobayashi T, Nishina Y, Tomoi H, Harada K, Tanaka K, Matsumoto E, Horimukai K, Ishihara J, Sasaki S, Inaba K, Seguchi K, Takahashi H, Salinas JL, Yamada Y. Corowa-kun: A messenger app chatbot delivers COVID-19 vaccine information, Japan 2021. Vaccine. 2022 Jul 30;40(32):4654-4662. doi: 10.1016/j.vaccine.2022.06.007. Epub 2022 Jun 8. PMID 35750541
- [Result] Weeks R, Cooper L, Sangha P, Sedoc J, White S, Toledo A, Gretz S, Lahav D, Martin N, Michel A, Lee JH, Slonim N, Bar-Zeev N. Chatbot-Delivered COVID-19 Vaccine Communication Message Preferences of Young Adults and Public Health Workers in Urban American Communities: Qualitative Study. J Med Internet Res. 2022 Jul 6;24(7):e38418. doi: 10.2196/38418. PMID 35737898
- [Result] 宋祎凡,刘晓雪,尹遵栋,等.2018-2020年中国9-45岁女性人乳头瘤病毒疫苗估算接种率[J].中国疫苗和免疫,2021,27(05):570-575.
- [Result] 邱丽蓉,牛战琴.9～14岁女性人乳头瘤病毒疫苗接种现状及其影响因素分析[J].中国生育健康杂志,2022,33(03):262-265.
- [Result] 史金晶,张肖肖,郑徽,等.中国大陆青少年家长人乳头瘤病毒疫苗认知度和接受度Meta分析[J].中国疫苗和免疫,2019,25(04):464-470.
- [Result] 武丽,马远珠,黄雪萍,等.广东省青少年女性对HPV疫苗知晓及接种意愿的调查研究[J].中国妇幼卫生杂志,2021,12(05):19-23.
- [Derived] Hou Z, Wu Z, Qu Z, Gong L, Peng H, Jit M, Larson HJ, Wu JT, Lin L. A vaccine chatbot intervention for parents to improve HPV vaccination uptake among middle school girls: a cluster randomized trial. Nat Med. 2025 Jun;31(6):1855-1862. doi: 10.1038/s41591-025-03618-6. Epub 2025 Apr 7. PMID 40195450
- See also: World Health Organization. Human papillomavirus vaccines: WHO position paper (2022 update). Weekly Epidemiological Record. 2022, 97 (50), 645-672. — https://www.who.int/publications/i/item/who-wer9750-645-672
- See also: World Health Organization. Behavioural and social drivers of vaccination: tools and practical guidance for achieving high uptake — https://www.who.int/publications/i/item/9789240049680